CLINICAL TRIAL: NCT01382420
Title: Long-term Effects of Adrenalectomy on Metabolic Syndrome, Glucose Metabolism, Lipid Metabolism, and Bone Metabolism in Subclinical Cushing's Syndrome of Adrenal Incidentaloma
Brief Title: Long-term Beneficial Metabolic Effects of Adrenalectomy in Subclinical Cushing's Syndrome of Adrenal Incidentaloma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Asan Medical Center (Other); Severance Hospital (Other); Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Jae Hyeon Kim, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-03-034
Record Dates: First submitted 2011-05-30; First posted 2011-06-27 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Cushing Syndrome
Keywords: subclinical cushing syndrome; hypercortisolism; adrenal incidentaloma; adrenalectomy
MeSH Terms: conditions — Cushing Syndrome; Adrenal incidentaloma | interventions — Surgical Procedures, Operative

ARMS (2):
- Adrenalectomy group (Active Comparator): patients who undergo adrenalectomy
  Interventions: Procedure: surgery
- Control group (No Intervention): patients who receive conservative treatment

INTERVENTIONS:
Procedure: surgery — adrenalectomy
  Arms: Adrenalectomy group

SUMMARY:
Objective:

To determine the metabolic effects of the adrenalectomy in subclinical Cushing's syndrome of adrenal incidentaloma.

Methods:

234 subclinical cushing syndrome and adrenal incidentaloma will be randomly assigned into two groups(e.g adrenalectomy group and conservative treatment group).

ELIGIBILITY:
Inclusion Criteria:

* patients with both unilateral adrenal incidentaloma and hypercortisolism
* definition of hypercortisolism

  * overnight dexamethasone suppression test, serum cortisol>1.8ug/dL
  * 24hr urine cortisol > upper reference limit

Exclusion Criteria:

* patients who took medication influencing cortisol secretion
* patients with definite clinical feature of cushing syndrome

  * moon face
  * abdominal striae
  * skin or proximal muscle atrophy
* metabolic syndrome, hyperthyroidism, hyperparathyroidism, chronic renal failure, rheumatic disease, hematologic disease
* patients who took following medication

  * insulin
  * oral hypoglycemic agent
  * thyroid hormone
  * anti-hyperlipidemic drug
  * sex hormone
* patients who taking steroid hormone or who took steroid hormone more than 2 weeks within 1 year
* psychiatric disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2011-05; Primary Completion 2020-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change of lipid profile between two groups | 4 Year
  lipid profile with LDL,apo B

SECONDARY OUTCOMES:
Incidence of obesity between two groups | 4Year
  measurement of body weight, height

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hyeon Kim, Study Director — Samsung Medical Center; Jung-Min Koh, Study Chair — M.D, Ph.D; Kee-Ho Song, Principal Investigator — M.D, Ph.D.; Yumie Rhee, Principal Investigator — M.D, Ph.D.
Locations (1):
- Samsung Medical Center, Seoul, South Korea